CLINICAL TRIAL: NCT02461160
Title: A Phase 1 Safety, Tolerability, Pharmacokinetic, Placebo-Controlled and Open-Label Study of Escalating Single and Multiple Oral Doses, Drug-Drug Interaction, Relative Bioavailability, Food Effect, and Effect on Elderly Subjects of TAK-915 in Healthy Subjects
Brief Title: Phase 1, TAK-915-1001, Single-Rising Dose, Multiple-Rising Dose, Drug-Drug Interaction, Relative Bioavailability, Food Effect, and Effect on Elderly Participants Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-915-1001; U1111-1168-6456 (Registry Identifier: WHO)
Record Dates: First submitted 2015-05-29; First posted 2015-06-03 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Midazolam; TAK-915

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (13):
- SRD Cohorts 1-3: Placebo (Placebo Comparator): TAK-915 placebo-matching suspension, orally, once on Day 1.
  Interventions: Drug: TAK-915 suspension
- SRD Cohort 1 TAK-915 30 mg (Experimental): TAK-915 30 mg suspension, orally, once on Day 1.
  Interventions: Drug: TAK-915 suspension
- SRD Cohort 2: TAK-915 100 mg (Experimental): TAK-915 100 mg suspension, orally, once on Day 1.
  Interventions: Drug: TAK-915 suspension
- SRD Cohort 3: TAK-915 200 mg (Experimental): TAK-915 200 mg suspension, orally, once on Day 1.
  Interventions: Drug: TAK-915 suspension
- MRD Cohorts 4-6 (Placebo Comparator): TAK-915 placebo-matching suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 placebo-matching suspension, orally, once on Days 8 to 14.
  Interventions: Drug: TAK-915 suspension
- MRD Cohort 4: TAK-915 30 mg (Experimental): TAK-915 30 mg suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 30 mg suspension, orally, once on Days 8 to 14.
  Interventions: Drug: TAK-915 suspension
- MRD Cohort 5: TAK-915 100 mg (Experimental): TAK-915 100 mg suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 100 mg suspension, orally, once on Days 8 to 14.
  Interventions: Drug: TAK-915 suspension
- MRD Cohort 6: TAK-915 200 mg (Experimental): TAK-915 200 mg suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 200 mg suspension, orally, once on Days 8 to 14.
  Interventions: Drug: TAK-915 suspension
- DDI Cohort 7: TAK-915 + Midazolam 2 mg (Experimental): Midazolam 2 mg suspension, orally, once on Day 1, followed by TAK-915 100 mg, suspension, orally, once on Day 3, followed by a 7-day washout period, followed by TAK-915 100 mg, suspension, orally, once, daily on Days 10 to 16 and Midazolam 2 mg solution, orally, once, on Day 16 (within 15 minutes after last dose of TAK-915).
  Interventions: Drug: TAK-915 suspension
- BA/FE Cohort 8 Group 1: A,B,C (Experimental): Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of Period 1, followed by Regimen B: TAK-915 50 mg, tablet, orally, under fasted conditions once on Day 1 of Period 2, followed by Regimen C: TAK-915 50 mg, tablet, orally under fed conditions once on Day 1 of Period 3. Each period was separated out by a 6 to 14-day washout period.
  Interventions: Drug: TAK-915 suspension
- BA/FE Cohort 9 Group 1: B,C,A (Experimental): Regimen B: TAK-915 50 mg, tablet, orally, under fasted conditions once on Day 1 of Period 2, followed by Regimen C: TAK-915 50 mg, tablet, orally under fed conditions once on Day 1 of Period 3 followed by Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of Period 1. Each period was separated out by a 6 to 14-day washout period.
  Interventions: Drug: TAK-915 suspension; Drug: Midazolam
- BA/FE Cohort 10 Group 1: C,A,B (Experimental): Regimen C: TAK-915 50 mg, tablet, orally under fed conditions once on Day 1 of Period 3 followed by Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of Period 1 followed by Regimen B: TAK-915 50 mg, tablet, orally, under fasted conditions once on Day 1 of Period 2. Each period was separated out by a 6 to 14-day washout period.
  Interventions: Drug: Placebo
- ESSD Cohort 11: TAK-915 50 mg (Experimental): TAK-915 50 mg, suspension, orally, under fasted conditions, once on Day 1 in participants aged 65 to 75 years.
  Interventions: Drug: TAK-915 suspension; Drug: TAK-915 tablet

INTERVENTIONS:
Drug: TAK-915 suspension — TAK-915 oral suspension
  Arms: BA/FE Cohort 8 Group 1: A,B,C; BA/FE Cohort 9 Group 1: B,C,A; DDI Cohort 7: TAK-915 + Midazolam 2 mg; ESSD Cohort 11: TAK-915 50 mg; MRD Cohort 4: TAK-915 30 mg; MRD Cohort 5: TAK-915 100 mg; MRD Cohort 6: TAK-915 200 mg; MRD Cohorts 4-6; SRD Cohort 1 TAK-915 30 mg; SRD Cohort 2: TAK-915 100 mg; SRD Cohort 3: TAK-915 200 mg; SRD Cohorts 1-3: Placebo
Drug: Midazolam — Midazolam oral solution
  Other Names: Versed
  Arms: BA/FE Cohort 9 Group 1: B,C,A
Drug: Placebo — Placebo-matching TAK-915 suspension
  Arms: BA/FE Cohort 10 Group 1: C,A,B
Drug: TAK-915 tablet — TAK-915 tablet
  Arms: ESSD Cohort 11: TAK-915 50 mg

SUMMARY:
The purpose of this study is to characterize the safety, tolerability and plasma pharmacokinetic (PK) profile of TAK-915 when administered as single and multiple oral suspension doses at escalating dose levels in healthy participants, including elderly participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-915. TAK-915 is being tested to find a safe and well-tolerated dose. This study will look at the pharmacokinetic characteristics (how the drug acts throughout the body) of the drug and safety and tolerability (lab results, vital signs, ECG, and side effects) in healthy people (including elderly) who take TAK-915.

The study will enroll a total of 88 patients. This study is designed to consist of 5 different dosing schedules: single rising dose (SRD), multiple rising dose (MRD), drug-drug interaction (DDI), bioavailability and food effect (BA/FE), and Elderly Subject Single Dose (ESSD). The study population for SRD will consist of 48 participants enrolled into 6 cohorts. Each cohort will have 8 randomized participants, with 6 receiving a single dose of TAK-915, and 2 receiving matching placebo under fasted conditions. The starting dose is 30 mg. The dose for Cohorts 2 through 6 will be determined based on data collected from previous cohorts.

The study population for MRD will consist of 32 participants enrolled into 4 cohorts. Each cohort will have 8 randomized participants, with 6 receiving one dose of TAK-915 on Day 1 and daily dosing on Days 8-14, and 2 receiving matching placebo under fasted conditions. The dose for each cohort in Part 2 will be determined based on data collected from completed SRD cohorts of the study.

The study population for DDI will consist of 12 participants enrolled into 1 cohort. All participants will receive one dose of TAK-915 on Day 3 and daily dosing on Days 10-16 under fasted conditions. All participants will also receive a single dose of Midazolam 2 mg on Day 1 and Day 16. The dose of TAK-915 in this cohort will be determined based on data collected from SRD cohorts and will be the same dose that is administered in MRD Cohort 8.

The study population for BA/FE will consist of 12 participants enrolled into 1 cohort. TAK-915 will be administered in 3 single-dose regimens in a 3-way crossover design using 50 mg oral dose treatments (Regimen A: TAK915 50 mg oral suspension formulation in fasted state; Regimen B: TAK-915 50 tablet formulation in fasted state; Regimen C: TAK-915 50 tablet formulation in fasted state). TAK-915 dosing will occur on Day 1 of each treatment period followed by a 14 day washout period.

The study population for ESSD will consist of 8 elderly participants (ages 65-75 years) enrolled into 1 cohort. All 8 participants will receive a single dose of TAK-915 50 mg suspension under fasted conditions.

This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 70 days. Participants will make multiple visits to the clinic including a period of confinement to the clinic and will be contacted by telephone 12 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy man or woman, aged 18 to 55 years, inclusive at the time of informed consent and first study medication dose for all cohorts will be included. Note that Cohort 12 will enroll healthy, elderly men and women, aged 65 to 75 years, inclusive.
4. Weighs at least 50 kg and has a body mass index (BMI) from 18.0 to 35.0 kg/m^2, inclusive at Screening.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
6. A female participant with no childbearing potential, defined as the participant has been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who are postmenopausal (defined as continuous amenorrhea of at least 2 y ears and follicle stimulating hormone (FSH) >40 IU/L).

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received TAK-915 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of TAK-915 and/or midazolam.
6. If female, the participant is of childbearing potential (eg. premenopausal, not sterilized).
7. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day 1).
8. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine.
9. Has taken any excluded medication, supplements, or food products during the time periods listed in the Excluded Medications and Dietary Products table.
10. Is pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study ; or intending to donate ova during such time period.
11. If male, the participant intends to donate sperm during the course of this study or for 12 weeks after the last dose of study medication.
12. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-915, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
13. Has mental retardation or medical condition that can cause cognitive impairment.
14. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
15. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Check-in (Day -1).
16. Has a positive test result for hepatitis B surface antigen (HBsAg), antibody to hepatitis C (anti -HCV) or a known history of human immunodeficiency virus infection at Screening.
17. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1). Cotinine test is positive at Screening or Check-in (Day -1).
18. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior the first dose of study medication.
19. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved and documented by signature by the principal investigator.
20. Has a supine blood pressure outside the ranges of 90 to 140 mmHg for systolic and 60 to 90 mmHg for diastolic, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
21. Has a resting heart rate outside the range 40 to 100 bpm, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
22. Has a QT interval with Fridericia correction method (QTcF) >430 ms (males) or >450 ms (females) or PR outside the range 120 to 220 ms, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
23. Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 the upper limits of normal.
24. Has a risk of suicide according to the Investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale [C-SSRS] or has made a suicide attempt in the previous 6 months).
25. Has poor peripheral venous access.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 12 May 2015 01 Aug 2016.
Pre-assignment Details: Healthy participants were enrolled to receive TAK-915 in any of the 5 parts of the study.
Groups:
- SRD Cohorts Pooled Placebo: TAK-915 placebo-matching suspension, orally, once on Day 1.
- MRD Cohorts Pooled Placebo: TAK-915 placebo-matching suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 placebo-matching suspension, orally, once on Days 8 to 14.
- MRD Cohort 5: TAK-915 30 mg: TAK-915 30 mg suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 30 mg suspension, orally, once on Days 8 to 14.
- MRD Cohort 6: TAK-915 100 mg: TAK-915 100 mg suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 100 mg suspension, orally, once on Days 8 to 14.
- MRD Cohort 7: TAK-915 200 mg: TAK-915 200 mg suspension, orally, once on Day 1, followed by a 7-day washout period, followed by TAK-915 200 mg suspension, orally, once on Days 8 to 14.
- DDI Cohort 8: TAK-915 + Midazolam 2 mg: Midazolam 2 mg suspension, orally, once on Day 1, followed by TAK-915 100 mg, suspension, orally, once on Day 3, followed by a 7-day washout period, followed by TAK-915 100 mg, suspension, orally, once, daily on Days 10 to 16 and Midazolam 2 mg solution, orally, once, on Day 16 (within 15 minutes after last dose of TAK-915).
- BA/FE Cohort 9 Group 1: A,B,C: Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of Period 1, followed by Regimen B: TAK-915 50 mg, tablet, orally, under fasted conditions once on Day 1 of Period 2, followed by Regimen C: TAK-915 50 mg, tablet, orally under fed conditions once on Day 1 of Period 3. Each period was separated out by a 6 to 14-day washout period.
- BA/FE Cohort 10 Group 2: B,C,A: Regimen B: TAK-915 50 mg, tablet, orally, under fasted conditions once on Day 1 of Period 2, followed by Regimen C: TAK-915 50 mg, tablet, orally under fed conditions once on Day 1 of Period 3 followed by Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of Period 1. Each period was separated out by a 6 to 14-day washout period.
- BA/FE Cohort 11 Group 3: C,A,B: Regimen C: TAK-915 50 mg, tablet, orally under fed conditions once on Day 1 of Period 3 followed by Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of Period 1 followed by Regimen B: TAK-915 50 mg, tablet, orally, under fasted conditions once on Day 1 of Period 2. Each period was separated out by a 6 to 14-day washout period.
- ESSD Cohort 12: TAK-915 50 mg: TAK-915 50 mg, suspension, orally, under fasted conditions, once on Day 1 in participants aged 65 to 75 years.
Period: Overall Study
Arm/Group | SRD Cohorts Pooled Placebo | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | MRD Cohorts Pooled Placebo | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | DDI Cohort 8: TAK-915 + Midazolam 2 mg | BA/FE Cohort 9 Group 1: A,B,C | BA/FE Cohort 10 Group 2: B,C,A | BA/FE Cohort 11 Group 3: C,A,B | ESSD Cohort 12: TAK-915 50 mg
Started | 8 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 12 | 4 | 4 | 4 | 8
Completed | 8 | 6 | 6 | 12 | 6 | 6 | 6 | 5 | 12 | 4 | 4 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SRD Cohorts Pooled Placebo | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | MRD Cohorts Pooled Placebo | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | DDI Cohort 8: TAK-915 + Midazolam 2 mg | BA/FE Cohort 9 Group 1: A,B,C | BA/FE Cohort 10 Group 2: B,C,A | BA/FE Cohort 11 Group 3: C,A,B | ESSD Cohort 12: TAK-915 50 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 12 | 4 | 4 | 4 | 8 | 88
Age, Continuous [Mean (Full Range); unit: Years] | 35.1 (9.76) [25 to 52] | 37.8 (16.68) [18 to 55] | 41.0 (12.47) [23 to 55] | 31.9 (6.76) [24 to 45] | 35.7 (11.36) [23 to 52] | 33.7 (4.32) [27 to 40] | 37.8 (5.74) [34 to 49] | 38.7 (10.03) [22 to 52] | 38.5 (8.53) [23 to 51] | 35.3 (14.36) [18 to 52] | 37.5 (12.34) [26 to 55] | 37.5 (8.70) [29 to 49] | 68.8 (2.25) [65 to 72] | 39.177 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 2 | 6 | 20
  Male | 7 | 5 | 4 | 10 | 6 | 6 | 5 | 5 | 10 | 2 | 4 | 2 | 2 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  Black or African American | 6 | 1 | 0 | 4 | 4 | 1 | 2 | 3 | 3 | 2 | 2 | 1 | 0 | 29
  White | 2 | 5 | 5 | 8 | 2 | 5 | 4 | 2 | 8 | 2 | 1 | 3 | 6 | 53
  Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or other Pacific islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 27.6 (4.41) [22 to 33] | 24.9 (5.26) [19 to 31] | 26.1 (2.95) [23 to 30] | 27.6 (3.99) [22 to 33] | 27.4 (1.71) [26 to 30] | 26.5 (3.00) [23 to 30] | 24.4 (3.95) [19 to 30] | 27.9 (2.52) [25 to 32] | 28.2 (2.23) [24 to 31] | 27.7 (6.33) [19 to 33] | 27.0 (1.52) [26 to 29] | 30.6 (2.93) [27 to 33] | 28.2 (2.75) [24 to 34] | 27.238 [19 to 34]
Smoking History [Number; unit: Participants]
  Particiapnt has never smoked | 6 | 5 | 6 | 11 | 5 | 5 | 4 | 4 | 10 | 4 | 3 | 3 | 7 | 73
  Particiapnt is a current smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Participant is an ex-smoker | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 14
Xanthine/caffeine history [Number; unit: Participants]
  Yes | 4 | 3 | 4 | 5 | 1 | 3 | 3 | 4 | 4 | 2 | 2 | 1 | 7 | 43
  No | 4 | 3 | 2 | 7 | 5 | 3 | 3 | 2 | 8 | 2 | 2 | 3 | 1 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 up to follow-up (SRD Cohorts: up to Day 13, MRD Cohorts: up to Day 26, DDI Cohort: up to Day 28, BA/FE Cohorts: up to Day 13, ESSD Cohort: up to Day 28)
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Groups:
- DDI Cohort 8: Midazolam 2 mg: Midazolam 2 mg suspension, orally, once on Days 1 and 16 (within 15 minutes after last dose of TAK-915).
- DDI Cohort 8: TAK-915 100 mg: TAK-915 100 mg, suspension, orally, once on Day 3, followed by a 7-day washout period, followed by TAK-915 100 mg, suspension, orally, once, daily on Days 10 to 16.
- BA/FE Cohort Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of ant period.
- BA/FE Cohort Regimen B: TAK-915 50 mg, tablet, orally, under fasted conditions once on Day 1 of any Period.
- BA/FE Cohort Regimen C: TAK-915 50 mg, tablet, orally under fed conditions once on Day 1 of any period.
Arm/Group | SRD Cohorts Pooled Placebo | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | MRD Cohorts Pooled Placebo | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | DDI Cohort 8: Midazolam 2 mg | DDI Cohort 8: TAK-915 100 mg | DDI Cohort 8: TAK-915 + Midazolam 2 mg | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 8 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 8
percentage of participants | 0 | 16.7 | 33.3 | 16.7 | 16.7 | 33.3 | 16.7 | 33.3 | 0 | 41.7 | 8.3 | 16.7 | 0 | 25 | 25

2. Primary Outcome: Percentage of Participants With Markedly Abnormal Safety Laboratory Tests
Description: The percentage of participants with any markedly abnormal standard safety laboratory values, including haematology, serum chemistries, or urinalysis, during the treatment period.
Time Frame: as for outcome 1
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SRD Cohorts Pooled Placebo | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | MRD Cohorts Pooled Placebo | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | DDI Cohort 8: Midazolam 2 mg | DDI Cohort 8: TAK-915 100 mg | DDI Cohort 8: TAK-915 + Midazolam 2 mg | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 8 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Measurements
Description: The percentage of participants who meet markedly abnormal criteria for vital signs after dosing, including oral body temperature (temp.), respiration rate, pulse rate (PR) Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) for assessment in positions of supine or standing. Vital signs were considered abnormal if they were beyond the values defined in categories.
Time Frame: as for outcome 1
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Groups:
- BA/FE Cohort Regimen A: TAK-915 50 mg, suspension, orally, under fasted conditions once on Day 1 of any period.
Arm/Group | SRD Cohorts Pooled Placebo | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | MRD Cohorts Pooled Placebo | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | DDI Cohort 8: Midazolam 2 mg | DDI Cohort 8: TAK-915 100 mg | DDI Cohort 8: TAK-915 + Midazolam 2 mg | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 8 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 8
percentage of participants
  Standing, after 1 minute SBP, <85 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 16.7 | 8.3 | 0 | 0 | 0 | 0
  Standing, after 1 minutes SBP, >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing, after 3 minutes SBP(mmHg), <85 mmHg | 0 | 0 | 0 | 8.3 | 0 | 0 | 16.7 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0
  Standing, after 3 minutes SBP, >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine, after 5 minutes SBP, <85 mmHg | 0 | 0 | 16.7 | 0 | 0 | 0 | 33.3 | 0 | 0 | 16.7 | 0 | 16.7 | 8.3 | 8.3 | 0
  Supine, after 5 minutes SBP, >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing, after 1 minute DBP, <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0 | 0 | 0 | 0
  Standing, after 1 minute DBP, >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing, after 3 minutes DBP, <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 8.3 | 0 | 0 | 0 | 0 | 0
  Standing, after 3 minutes DBP, >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine, after 5 minutes DBP, <50 mmHg | 12.5 | 0 | 16.7 | 8.3 | 0 | 0 | 33.3 | 0 | 8.3 | 0 | 8.3 | 8.3 | 0 | 0 | 12.5
  Supine, after 5 minutes DBP, >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing, after 1 min PR, <50 beats/min | 0 | 0 | 0 | 0 | 33.3 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing, after 1 min PR, >120 beats/min | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 33.3 | 0 | 8.3 | 0 | 0 | 0 | 8.3 | 0
  Standing, after 3 mins PR, <50 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 8.3 | 0 | 0 | 0 | 0
  Standing, after 3 mins PR, >120 beats/min | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 16.7 | 16.7 | 0 | 8.3 | 8.3 | 8.3 | 0 | 0 | 0
  Supine, after 5 mins PR, <50 beats/min | 25 | 0 | 16.7 | 16.7 | 50 | 50 | 50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine, after 5 mins PR, >120 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing, after 1 min Temperature, <35.6 °C | 0 | 16.7 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  Standing, after 1 min Temperature, >37.7 °C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing, after 3 mins Temperature, <35.6 °C | 0 | 16.7 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  Standing, after 3 mins Temperature, >37.7 °C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine, after 5 mins Temperature, <35.6 °C | 0 | 16.7 | 0 | 16.7 | 16.7 | 33.3 | 0 | 16.7 | 0 | 8.3 | 0 | 0 | 0 | 8.3 | 12.5
  Supine, after 5 mins Temperature, >37.7 °C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With Markedly Abnormal Values of 12-Lead Electrocardiogram (ECG) Parameters
Description: The percentage of participants who meet markedly abnormal criteria for ECG parameters as specified by the protocol and statistical analysis plan during the treatment period. ECG parameters were considered abnormal if they were beyond the values defined in categories.
Time Frame: as for outcome 1
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SRD Cohorts Pooled Placebo | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | MRD Cohorts Pooled Placebo | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | DDI Cohort 8: Midazolam 2 mg | DDI Cohort 8: TAK-915 100 mg | DDI Cohort 8: TAK-915 + Midazolam 2 mg | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 8 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 8
percentage of participants
  Heart Rate, <50 beats/min | 37.5 | 0 | 16.7 | 25 | 66.7 | 50 | 50 | 0 | 0 | 0 | 0 | 8.3 | 0 | 0 | 0
  Heart Rate, >120 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval, <=80 msec (ms) | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval, >=200 ms | 12.5 | 16.7 | 0 | 8.3 | 33.3 | 16.7 | 16.7 | 33.3 | 8.3 | 8.3 | 16.7 | 25 | 25 | 8.3 | 12.5
  QRS Interval, <=80 ms | 12.5 | 16.7 | 16.7 | 8.3 | 0 | 0 | 0 | 33.3 | 8.3 | 25.0 | 25.0 | 16.7 | 16.7 | 8.3 | 25
  QRS Interval, >=180 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval, <=300 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval, >=460 ms | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5
  QTcB Interval, <=300 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval,≥500ms OR ≥450ms and ≥30ms CFB | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 8.3 | 0 | 0
  QTcF Interval, <= 300 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, ≥500 msec OR ≥ 450 msec and ≥30 CFB | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-915
Time Frame: SRD and ESSD Cohorts: Day 1 pre-dose and at multiple timepoints (up to 96 hours) post dose; MRD cohorts: Days 1, 8 and 14 pre-dose and at multiple timepoints (up to 96 hours) post dose
Population: Pharmacokinetic set included all participants who received study drug and have at least 1 measurable plasma concentration or amount of drug in the urine for either TAK-915 or its metabolite M-I or for midazolam or its metabolite 1-hydroxymidazolam.
Measure: Median (Full Range); unit: hr
Groups:
- SRD Cohort 4: TAK-915 200 mg: TAK-915 200 mg suspension, orally via syringe, once on Day 1.
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
hr
  Day 1 | 1.750 [1.50 to 6.00] | 2.000 [0.50 to 4.00] | 2.000 [1.00 to 3.00] | 2.508 [1.00 to 6.10] | 1.500 [1.50 to 3.00] | 1.500 [1.00 to 4.00] | 3.058 [3.00 to 6.00] | 1.500 [1.00 to 2.00]
  Day 8 | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | 1.500 [1.50 to 2.00] | 2.000 [1.50 to 4.00] | 2.00 [1.50 to 3.00] | NA [NA to NA] — Data was not analysed for this arm group at the given time point.
  Day 14 | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | NA [NA to NA] — Data was not analysed for this arm group at the given time point. | 1.500 [1.50 to 1.52] | 2.500 [1.00 to 4.00] | 3.000 [1.00 to 4.00] | NA [NA to NA] — Data was not analysed for this arm group at the given time point.

6. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-915
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
ng/mL
  Day 1 | 203.7 (42.77) [1.50 to 6.00] | 654.8 (145.97) [0.50 to 4.00] | 417.3 (96.27) [1.00 to 3.00] | 675.8 (168.66) [1.00 to 6.10] | 209.5 (46.60) [1.50 to 3.00] | 651.8 (227.77) [1.00 to 4.00] | 743.8 (148.45) [3.00 to 6.00] | 414.0 (106.43) [1.00 to 2.00]
  Day 8 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 196.0 (47.72) [1.50 to 2.00] | 651.0 (130.51) [1.50 to 4.00] | 836.7 (220.01) [1.50 to 3.00] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 397.5 (137.14) [1.50 to 1.52] | 1081.0 (170.94) [1.00 to 4.00] | 1865.0 (334.71) [1.00 to 4.00] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.

7. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for TAK-915
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
ng*hr/mL
  Day 1 | 2560.0 (631.76) [1.50 to 6.00] | 8293.3 (1430.62) [0.50 to 4.00] | 5478.1 (729.80) [1.00 to 3.00] | 10285.1 (1515.01) [1.00 to 6.10] | 2610.0 (534.55) [1.50 to 3.00] | 7984.6 (1437.41) [1.00 to 4.00] | 11640.5 (1889.06) [3.00 to 6.00] | 4693.0 (637.27) [1.00 to 2.00]
  Day 8 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 2301.7 (782.55) [1.50 to 2.00] | 8333.9 (890.57) [1.50 to 4.00] | 12549.3 (3355.02) [1.50 to 3.00] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 5688.9 (2759.15) [1.50 to 1.52] | 15068.7 (2367.02) [1.00 to 4.00] | 31656.0 (5574.82) [1.00 to 4.00] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.

8. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-915
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
ng*hr/mL
  Day 1 | 5187.3 (956.99) | 18229.5 (5124.97) | 10812.4 (1098.50) | 24204.7 (3870.08) | 5380.9 (2065.75) | 15640.0 (2998.50) | 30251.6 (4473.58) | 11552.2 (2214.35)
  Day 8 | NA (NA) — Data was not analysed for this arm group at the given time point. | NA (NA) — Data was not analysed for this arm group at the given time point. | NA (NA) — Data was not analysed for this arm group at the given time point. | NA (NA) — Data was not analysed for this arm group at the given time point. | 2301.7 (782.55) | 8334.6 (890.88) | 12549.3 (3355.02) | NA (NA) — Data was not analysed for this arm group at the given time point.
  Day 14 | NA (NA) — Data was not analysed for this arm group at the given time point. | NA (NA) — Data was not analysed for this arm group at the given time point. | NA (NA) — Data was not analysed for this arm group at the given time point. | NA (NA) — Data was not analysed for this arm group at the given time point. | 12653.2 (8536.11) | 27924.7 (7330.59) | 67706.4 (22451.23) | NA (NA) — Data was not analysed for this arm group at the given time point.

9. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-915
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
ng*hr/mL | 6197.1 (1102.70) [1.50 to 6.00] | 19345.6 (5548.95) [0.50 to 4.00] | 12198.3 (1312.58) [1.00 to 3.00] | 30243.3 (7208.93) [1.00 to 6.10] | 6565.6 (3237.81) [1.50 to 3.00] | 17507.2 (4461.40) [1.00 to 4.00] | 40326.7 (11260.16) [3.00 to 6.00] | 16991.5 (4349.17) [1.00 to 2.00]

10. Primary Outcome: Rac(AUC): Accumulation Ratios Between Day 14 AUC(0-24) and Day 1 AUC(0-24) for TAK-915
Time Frame: Days 1 and 14 pre-dose and at multiple time points (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 2.100 (0.6568) | 1.973 (0.6523) | 2.761 (0.5207)

11. Primary Outcome: Rac(Cmax): Accumulation Ratios Between Day 14 Cmax and Day 1 Cmax for TAK-915
Time Frame: Days 1 and 14 pre-dose and at multiple time points (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 1.884 (0.4627) | 1.859 (0.7642) | 2.556 (0.5148)

12. Primary Outcome: Time Dependency Assessment From AUC(0-24) After Last Dose for TAK-915 on Day 14 in MRD Cohorts Compared to AUC(0-inf) After a Single Dose on Day 1
Time Frame: Days 1 and 14 pre-dose and at multiple time points (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio | 0.873 (0.1342) | 0.883 (0.1441) | 0.846 (0.1463)

13. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Midazolam Alone (Day 1) and in the Presence of TAK-915 (Day 16) in DDI Cohort
Time Frame: Days 1 and 16 pre-dose and at multiple timepoints (up to 24 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DDI Cohort 7: TAK-915 + Midazolam 2 mg
Number analyzed (Participants) | 6
ng/mL
  Day 1 | 9.6 (3.02)
  Day 16 | 8.3 (2.17)

14. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for Midazolam Alone (Day 1) and in the Presence of TAK-915 (Day 16) in DDI Cohort
Time Frame: Days 1 and 16 pre-dose and at multiple timepoints (up to 24 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | DDI Cohort 7: TAK-915 + Midazolam 2 mg
Number analyzed (Participants) | 12
ng*hr/mL
  Day 1 | 25.0 (10.09)
  Day 16 | 17.4 (5.48)

15. Primary Outcome: AUC(0-24) for Midazolam After Single Dose (Day 1)/AUC(0-24) for Midazolam After 7 Daily Doses of TAK-915 (Day 16) in DDI Cohort
Time Frame: Days 1 and 16 pre-dose and at multiple timepoints (up to 24 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | DDI Cohort 7: TAK-915 + Midazolam 2 mg
Number analyzed (Participants) | 12
Ratio | 0.735 (0.1509)

16. Secondary Outcome: Terminal Elimination Half-life (t1/2) for TAK-915
Time Frame: SRD and ESSD Cohorts: Day 1 pre-dose and at multiple timepoints (up to 96 hours) post dose; MRD cohorts: Days 1 and 14 pre-dose and at multiple timepoints (up to 96 hours) post dose
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
hr
  Day 1 | 35.246 (42.77) [22.74 to 55.60] | 34.008 (145.97) [27.05 to 85.65] | 32.621 (96.27) [23.02 to 39.02] | 37.826 (168.66) [29.50 to 55.78] | 37.166 (46.60) [20.08 to 50.02] | 23.326 (227.77) [18.77 to 46.44] | 46.408 (148.45) [24.33 to 78.31] | 61.244 (106.43) [27.71 to 75.78]
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 32.770 (137.14) [22.97 to 61.40] | 23.517 (170.94) [17.57 to 28.73] | 35.503 (334.71) [24.75 to 54.51] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.

17. Secondary Outcome: CL/F: Apparent Clearance for TAK-915
Time Frame: as for outcome 16
Population: Pharmacokinetic set included all participants who received study drug and have at least 1 measurable plasma concentration or amount of drug in the urine for either TAK-915 or its metabolite M-I or for midazolam or its metabolite 1-hydroxymidazolam. Number of participants analysed is the participants who were evaluable in each cohort.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 8
L/hr
  Day 1 | 4.966 (0.8498) [22.74 to 55.60] | 5.565 (1.7418) [27.05 to 85.65] | 16.566 (1.9026) [23.02 to 39.02] | 6.928 (1.5930) [29.50 to 55.78] | 5.437 (2.3306) [20.08 to 50.02] | 5.993 (1.3303) [18.77 to 46.44] | 5.313 (1.6232) [24.33 to 78.31] | 5.651 (2.3825) [27.71 to 75.78]
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 6.289 (2.6024) [22.97 to 61.40] | 6.791 (1.1948) [17.57 to 28.73] | 6.625 (1.2982) [24.75 to 54.51] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.

18. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for TAK-915
Time Frame: as for outcome 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
L
  Day 1 | 271.621 (81.4842) [22.74 to 55.60] | 253.274 (44.1565) [27.05 to 85.65] | 739.900 (138.9342) [23.02 to 39.02] | 384.373 (54.7107) [29.50 to 55.78] | 253.191 (43.9653) [20.08 to 50.02] | 219.807 (44.0421) [18.77 to 46.44] | 289.052 (33.6825) [24.33 to 78.31] | 251.206 (28.7250) [27.71 to 75.78]
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 290.034 (47.4883) [22.97 to 61.40] | 231.463 (38.5789) [17.57 to 28.73] | 373.816 (143.239) [24.75 to 54.51] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.

19. Secondary Outcome: Total Amount of Drug Excreted in Urine (Ae) for TAK-915
Time Frame: SRD Cohorts: Day 1 pre-dose and at multiple timepoints (up to 96 hours) post dose; MRD cohorts: Days 1 and 14 pre-dose and at multiple timepoints (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng
  Day 1 | 10716.238 (6732.8265) [22.74 to 55.60] | 56307.372 (22847.5616) [27.05 to 85.65] | 39016.323 (39432.2098) [23.02 to 39.02] | 70789.157 (31812.6780) [29.50 to 55.78] | 11637.538 (7559.7833) [20.08 to 50.02] | 75873.405 (57990.3620) [18.77 to 46.44] | 84953.950 (28044.2529) [24.33 to 78.31]
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 23712.223 (16960.3220) [22.97 to 61.40] | 107635.360 (66665.1502) [17.57 to 28.73] | 173279.223 (102551.0702) [24.75 to 54.51]

20. Secondary Outcome: Fraction of Drug Excreted in Urine (Fe) for TAK-915
Time Frame: as for outcome 19
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: fraction excreted
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
fraction excreted
  Day 1 | 0.036 (0.0224) [22.74 to 55.60] | 0.056 (0.0228) [27.05 to 85.65] | 0.020 (0.0197) [23.02 to 39.02] | 0.035 (0.0159) [29.50 to 55.78] | 0.039 (0.0252) [20.08 to 50.02] | 0.076 (0.0580) [18.77 to 46.44] | 0.042 (0.0140) [24.33 to 78.31]
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 0.079 (0.0565) [22.97 to 61.40] | 0.108 (0.0667) [17.57 to 28.73] | 0.099 (0.0471) [24.75 to 54.51]

21. Secondary Outcome: Renal Clearance (CLr) for TAK-915
Time Frame: as for outcome 19
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/hr
  Day 1 | 2.140 (1.3783) [22.74 to 55.60] | 3.191 (1.1645) [27.05 to 85.65] | 3.612 (3.5780) [23.02 to 39.02] | 2.915 (1.3632) [29.50 to 55.78] | 2.265 (1.7248) [20.08 to 50.02] | 5.047 (4.2166) [18.77 to 46.44] | 2.934 (1.2499) [24.33 to 78.31]
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 2.208 (0.8706) [22.97 to 61.40] | 4.696 (4.5467) [17.57 to 28.73] | 3.246 (2.0065) [24.75 to 54.51]

22. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-915 on Day 1 in DDI Cohort
Time Frame: Days 1 at multiple time points (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DDI Cohort 7: TAK-915 + Midazolam 2 mg
Number analyzed (Participants) | 12
ng/mL | 519.7 (156.12)

23. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for TAK-915 on Day 1 in DDI Cohort
Time Frame: Days 1 at multiple time points (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | DDI Cohort 7: TAK-915 + Midazolam 2 mg
Number analyzed (Participants) | 12
ng*hr/mL | 7324.5 (2130.73)

24. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-Time Curve From Time 0 to Time Tau Over a Dosing Interval Where Tau is the Length of the Dosing Interval for TAK-915 in DDI Cohort
Time Frame: Days 16 at multiple time points (up to 96 hours) post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | DDI Cohort 7: TAK-915 + Midazolam 2 mg
Number analyzed (Participants) | 12
ng*hr/mL | 17093.9 (5803.03)

25. Secondary Outcome: Ratio of TAK-915 Metabolite Cmax to TAK-915 Cmax in SRD and MRD Cohorts
Time Frame: Day 1 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8
ratio
  Day 1 | 0.230 (0.0281) [22.74 to 55.60] | 0.248 (0.0440) [27.05 to 85.65] | 0.254 (0.0287) [23.02 to 39.02] | 0.273 (0.0550) [29.50 to 55.78] | 0.212 (0.0410) [20.08 to 50.02] | 0.267 (0.0454) [18.77 to 46.44] | 0.277 (0.0632) [24.33 to 78.31] | 0.207 (0.0326) [27.71 to 75.78]
  Day 14 | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point. | 0.356 (0.0609) [22.97 to 61.40] | 0.480 (0.0764) [17.57 to 28.73] | 0.0764 (0.0690) [24.75 to 54.51] | NA (NA) [NA to NA] — Data was not analysed for this arm group at the given time point.

26. Secondary Outcome: Ratio of TAK-915 Metabolite AUC(0-inf) to TAK-915 AUC(0-inf) in SRD Cohorts
Time Frame: Day 1 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | SRD Cohort 4: TAK-915 200 mg | ESSD Cohort 12: TAK-915 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
ratio | 0.492 (0.1179) [22.74 to 55.60] | 0.475 (0.1029) [27.05 to 85.65] | 0.483 (0.1037) [23.02 to 39.02] | 0.576 (0.1071) [29.50 to 55.78] | 0.451 (0.1334) [27.71 to 75.78]

27. Secondary Outcome: Ratio of TAK-915 Metabolite Area Under the Plasma Concentration-Time Curve From Time 0 to Time Tau Over a Dosing Interval [AUC(0-tau)] Where Tau is the Length of the Dosing Interval to TAK-915 AUC(0-tau) in MRD Cohorts
Time Frame: Day 14 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio | 0.496 (0.1177) [20.08 to 50.02] | 0.640 (0.1177) [18.77 to 46.44] | 0.505 (0.0940) [24.33 to 78.31]

28. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-915 and TAK-915 Metabolite M-I in BA/FE Cohort
Time Frame: Day 1 of Periods 1, 2 and 3 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C
Number analyzed (Participants) | 12 | 12 | 12
ng/mL
  TAK-915 | 337.0 (337.0) | 208.0 (68.48) | 143.4 (55.03)
  Metabolite M-I | 79.2 (18.55) | 48.9 (13.21) | 34.6 (16.03)

29. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-915 and TAK-915 Metabolite M-I in BA/FE Cohort
Time Frame: Day 1 of Periods 1, 2 and 3 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C
Number analyzed (Participants) | 12 | 12 | 12
ng*hr/mL
  TAK-915 | 8412.3 (2019.40) | 7310.0 (1928.95) | 5740.2 (2227.13)
  Metabolite M-I | 3785.3 (771.24) | 2992.1 (582.21) | 2208.7 (888.83)

30. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-915 and TAK-915 Metabolite M-I in BA/FE Cohort
Time Frame: Day 1 of Periods 1, 2 and 3 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C
Number analyzed (Participants) | 12 | 12 | 12
ng*hr/mL
  TAK-915 | 10155.2 (2909.10) | 9414.5 (9414.5) | 7151.5 (2836.73)
  Metabolite M-I | 4727.2 (1073.11) | 4145.2 (1027.33) | 3011.6 (1315.23)

31. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-915 and TAK-915 Metabolite M-I in BA/FE Cohort
Time Frame: Day 1 of Periods 1, 2 and 3 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C
Number analyzed (Participants) | 12 | 12 | 12
hr
  TAK-915 | 1.500 [1.00 to 3.40] | 3.000 [1.50 to 6.00] | 7.000 [4.08 to 24.00]
  Metabolite M-I | 2.250 [1.00 to 12.00] | 10.000 [2.00 to 24.00] | 24.000 [10.00 to 32.00]

32. Secondary Outcome: Terminal Elimination Half-life (t1/2) for TAK-915 and TAK-915 Metabolite M-I in BA/FE Cohort
Time Frame: Day 1 of Periods 1, 2 and 3 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C
Number analyzed (Participants) | 12 | 12 | 12
hr
  TAK-915 | 34.973 [19.83 to 52.65] | 45.359 [21.43 to 63.71] | 40.101 [19.46 to 53.53]
  Metabolite M-I | 39.937 [19.68 to 68.78] | 50.010 [19.55 to 142.18] | 48.406 [19.43 to 76.85]

33. Secondary Outcome: λz: Terminal Elimination Rate Constant for TAK-915 and TAK-915 Metabolite M-I in BA/FE Cohort
Time Frame: Day 1 of Periods 1, 2 and 3 predose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C
Number analyzed (Participants) | 12 | 12 | 12
1/hr
  TAK-915 | 0.0202 (0.00623) | 0.0187 (0.00677) | 0.0202 (0.00702)
  Metabolite M-I | 0.0180 (0.00665) | 0.0155 (0.00834) | 0.0162 (0.00748)

ADVERSE EVENTS:
Time Frame: Day 1 up to follow-up (SRD Cohorts: up to Day 13, MRD Cohorts: up to Day 26, DDI Cohort: up to Day 28, BA/FE Cohorts: up to Day 13, ESSD Cohort: up to Day 28)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Adverse events were summarized as per the regimen received by the participants.
Arm/Group | SRD Cohorts Pooled Placebo | SRD Cohort 1 TAK-915 30 mg | SRD Cohort 2: TAK-915 100 mg | SRD Cohort 3: TAK-915 200 mg | MRD Cohorts Pooled Placebo | MRD Cohort 5: TAK-915 30 mg | MRD Cohort 6: TAK-915 100 mg | MRD Cohort 7: TAK-915 200 mg | DDI Cohort 8: Midazolam 2 mg | DDI Cohort 8: TAK-915 100 mg | DDI Cohort 8: TAK-915 + Midazolam 2 mg | BA/FE Cohort Regimen A | BA/FE Cohort Regimen B | BA/FE Cohort Regimen C | ESSD Cohort 12: TAK-915 50 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 1/6 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/6 | 2/6 | 2/12 | 1/6 | 2/6 | 1/6 | 1/6 | 0/12 | 5/12 | 1/12 | 2/12 | 0/12 | 3/12 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRD Cohorts Pooled Placebo (N=8) | SRD Cohort 1 TAK-915 30 mg (N=6) | SRD Cohort 2: TAK-915 100 mg (N=6) | SRD Cohort 3: TAK-915 200 mg (N=12) | MRD Cohorts Pooled Placebo (N=6) | MRD Cohort 5: TAK-915 30 mg (N=6) | MRD Cohort 6: TAK-915 100 mg (N=6) | MRD Cohort 7: TAK-915 200 mg (N=6) | DDI Cohort 8: Midazolam 2 mg (N=12) | DDI Cohort 8: TAK-915 100 mg (N=12) | DDI Cohort 8: TAK-915 + Midazolam 2 mg (N=12) | BA/FE Cohort Regimen A (N=12) | BA/FE Cohort Regimen B (N=12) | BA/FE Cohort Regimen C (N=12) | ESSD Cohort 12: TAK-915 50 mg (N=8)
Anxiety (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRD Cohorts Pooled Placebo (N=8) | SRD Cohort 1 TAK-915 30 mg (N=6) | SRD Cohort 2: TAK-915 100 mg (N=6) | SRD Cohort 3: TAK-915 200 mg (N=12) | MRD Cohorts Pooled Placebo (N=6) | MRD Cohort 5: TAK-915 30 mg (N=6) | MRD Cohort 6: TAK-915 100 mg (N=6) | MRD Cohort 7: TAK-915 200 mg (N=6) | DDI Cohort 8: Midazolam 2 mg (N=12) | DDI Cohort 8: TAK-915 100 mg (N=12) | DDI Cohort 8: TAK-915 + Midazolam 2 mg (N=12) | BA/FE Cohort Regimen A (N=12) | BA/FE Cohort Regimen B (N=12) | BA/FE Cohort Regimen C (N=12) | ESSD Cohort 12: TAK-915 50 mg (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.